CLINICAL TRIAL: NCT06753643
Title: Implementing the National Frailty Policy in Singapore's Primary Care: A Pilot Feasibility Study of The Intrinsic Capacity ProMotion in PrimAry Care for The Frail Program (IMPACTFrail)
Brief Title: An Intrinsic Capacity Identification and Management Programme for Older Adults in Singapore's Primary Care
Acronym: IMPACTFrail
Status: Not yet recruiting | Type: Observational
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: National Healthcare Group Polyclinics (Other Government); National University Polyclinics (Unknown); SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Other Study IDs: GERI1637
Record Dates: First submitted 2024-12-11; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Healthy Ageing; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults (programme recipients): These are the recipients of the new programme in this feasibility study.
  Main study components of direct involvement. Qualitative - Focus group discussions or in-depth interviews with programme recipients
  Quantitative - Monitoring process indicators
  Interventions: Other: The IMPACTFrail programme

INTERVENTIONS:
Other: The IMPACTFrail programme — The IMPACTFrail programme

SUMMARY:
The IMPACTFrail program is an intrinsic capacity (IC) identification and management program for mildly frail older adults. Specifically, it delivers the three-tier approach recommended in the National Frailty Strategy Policy Report. The program's core functions include the segmentation of older persons using the Clinical Frailty Scale (CFS) score followed by secondary IC screening for CFS 4 to 5 (Tier 1), follow-up clinical assessment to confirm IC losses (Tier 2) and needs-directed management and tracking of their health (Tier 3).

The investigator aims to conduct a multi-site feasibility study on a small group of older adult study participants (n=30 per polyclinic).

The feasibility study has a few components. First, a qualitative study will assess its feasibility (implementation, appropriateness, acceptability, practicality, adaptability) as perceived by older adults, healthcare providers, and healthcare administrators. Second, the investigator aims to collect process indicators to track its implementation progress. Third, program costs will be estimated. Fourth, the investigator will develop a logic model and theory of change, and cluster-specific detailed written program descriptions. Lastly, the investigator aims to triangulate the findings and assess the feasibility for larger-scale implementation. This study is guided by implementation science frameworks and guidelines for conducting feasibility studies.

DETAILED DESCRIPTION:
Background:

The broad goal for older adults is to age well and have healthy ageing. WHO defines healthy ageing as "the process of developing and maintaining the functional ability that enables wellbeing in older age." Functional ability is about having the capabilities that enable all people to be and do what they have reason to value.

Frailty is a clinically recognisable state whereby an older person's ability to cope with daily or acute stressors is compromised as a result of vulnerability from age-related deterioration in physiological reserves and function across multiple organ systems. Frailty is associated with negative health outcomes and is expected to increase in Singapore's ageing population. The National Frailty Strategy Policy Report published in 2023 serves to guide the Singapore Ministry of Health (MOH) Frailty Policy Implementation Workgroup in implementing the National Frailty Policy (NFP). One of the gaps identified in the report was the need for coordinated care and continuity of care across health and social service providers for frail older adults. To address this gap in Singapore's primary care setting, the IMPACTFrail program's core functions are to conduct segmentation of older people by using the Clinical Frailty Scale (CFS) score followed by secondary intrinsic capacity (IC) screening of six domains (locomotion, vision, hearing, vitality, cognition, psychological capacity) for CFS 4 and 5 (Tier 1), follow-up assessments based on IC deficits detected at screening (Tier 2), and coordination, management, and tracking (Tier 3). This study aims to co-develop IMPACTFrail's intervention components and implementation strategies in a small number of polyclinics and test its feasibility using implementation research in real-world local contexts.

Methods:

Prior to this pilot feasibility study, the investigators co-developed the innovation and implementation strategies among GERI, polyclinic cluster representatives, and implementers. This will be guided by the UK Medical Research Council's Framework (MRC) for developing and evaluating complex interventions and Framework of Actions for Intervention Development (FAID). Informal FGDs and interviews with stakeholders were conducted and the findings used to inform the development of the innovation. ERIC strategies will be selected to address CFIR barriers identified from the FGDs/interviews and specify and develop them.

Here, the investigators aim to conduct a multi-site feasibility study, with a few components. Each polyclinic has highly contextualised barriers, workflows, and infrastructure. Thus, each polyclinic is conceptualised as a single site for feasibility testing. There is no comparator arm.

First, FGDs/IDIs will be conducted to assess the program's feasibility (implementation, acceptability, practicality, adaptability) as perceived by older adults, healthcare providers, and healthcare administrators.

Second, the investigators aim to collect process indicators to track the program's implementation progress.

Third, program costs will be estimated.

Fourth, the investigators will develop a logic model and theory of change, and cluster-specific detailed written program descriptions.

Lastly, the investigators aim to triangulate our findings and assess the feasibility for larger-scale implementation.

This study is guided by implementation science frameworks and guidelines for conducting feasibility studies.

Discussion:

This project aims to improve the lives of older people through early detection and management of IC deficits for those with mild frailty (CFS 4-5) in primary care. This promotes longer-term outcomes including functional ability, improved quality of life, reduced healthcare use, and lower mortality.

Additionally:

First, the project translates evidence on the optimisation of IC and functional ability for healthy ageing to practice and policy in Singapore's primary care. Second, there is knowledge creation. This study contributes to the local evidence on screening and management strategies for delaying frailty progression by addressing IC deficits in frail older persons. The investigators inform the adaptations to implement the WHO ICOPE framework in local primary care contexts. Additionally, the project contributes to a better understanding on the optimisation of resources to groups who may benefit the most, by targeting CFS 4 and 5 for IC screening and delivering resource-intensive assessment and downstream interventions to this subgroup. Third, this study involves engaging all three clusters from the outset to accelerate national-level implementation and scaling up.

Additionally, to increase the likelihood of scalability, the investigators will involve 3 clusters and 1-2 polyclinics from each cluster. Fourth, the study offers opportunities for knowledge exchange.

Lastly, the project is aligned with national strategies like HealthierSG (informs frailty protocols for management in primary care), Age Well SG (enables frail community-dwelling persons to age in place), and the 2023 Action Plan for Successful Ageing (optimising IC and functional ability through a health program).

ELIGIBILITY:
Older Adults

Inclusion Criteria:

* being a patient of the polyclinic site
* aged 60 years and above
* Clinical frailty score (CFS) of 4 - 5
* Not done comprehensive geriatric assessment (CGA) in the past 12 months (based on available medical records or self-report)
* Not a current patient of geriatric specialist outpatient clinic (based on available medical records or self-report).

Exclusion Criteria:

* Do not meet inclusion criteria above

Healthcare Staff (for qualitative study)

Inclusion Criteria:

* aged 21 years and above
* Involved in the IMPACTFrail program as an implementer and/or a healthcare administrator with authority to make implementation decisions.

Exclusion Criteria:

* Do not meet inclusion criteria above

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults will be polyclinic patients aged 60 years and above with CFS score 4 or 5 as assigned by a trained healthcare provider at the polyclinic. They should not have done any comprehensive geriatric assessment or be currently receiving geriatric specialist outpatient services.
  Healthcare staff can be polyclinic healthcare providers (e.g., polyclinic doctors, nurses, care coordinators, care managers, medical social workers). Healthcare administrators would be from the polyclinic leadership team, who are decision-makers who have the authority to make implementation decisions and are familiar with the overall frailty and IC management strategies in primary care in Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Qualitative study 1 | Mar 2025 - Feb 2026
  What will be measured:
  Deviations to the intended execution of the programme and implementation strategies and reasons for changes made.
  How will it be measured:
  Via in-depth interviews (IDIs) and focus group discussions (FGDs) with healthcare administrators and healthcare providers.
  All participants for the qualitative study will be identified through purposive sampling. We will adopt the Rapid Qualitative Inquiry (RQI) approach in data analysis.
Qualitative study 2 | Mar 2025 - Feb 2026
  What will be measured:
  Barriers/facilitators of implementing/receiving the programme and its implementation strategies.
  How will it be measured:
  Via in-depth interviews (IDIs) and focus group discussions (FGDs) with healthcare administrators, healthcare providers, and older adults.
  All participants for the qualitative study will be identified through purposive sampling. We will adopt the Rapid Qualitative Inquiry (RQI) approach in data analysis.
Qualitative study 3 | Mar 2025 - Feb 2026
  What will be measured:
  Perspectives on the ability to deliver innovation with given resources (manpower, infrastructure, IT, others).
  How will it be measured:
  Via in-depth interviews (IDIs) and focus group discussions (FGDs) with healthcare administrators and healthcare providers.
  All participants for the qualitative study will be identified through purposive sampling. We will adopt the Rapid Qualitative Inquiry (RQI) approach in data analysis.
Qualitative study 4 | Mar 2025 - Feb 2026
  What will be measured:
  Suggestions on how to improve the implementation of the programme for scalability and sustainability.
  How will it be measured:
  Via in-depth interviews (IDIs) and focus group discussions (FGDs) with healthcare administrators and healthcare providers.
  All participants for the qualitative study will be identified through purposive sampling. We will adopt the Rapid Qualitative Inquiry (RQI) approach in data analysis.
Programme cost | Mar 2025 - Feb 2026
  The aim is to inform the funding of resources (developmental cost e.g., training, new materials, innovation cost and cost of implementation strategies needed to scale up the programme).
  Programme costs will be derived by aggregating expenditures from financial statements on operating expenses, manpower, training, and equipment cost incurred, and obtaining the time spent by healthcare workers to actualise the delivery of the program.
Logic model and theory of change | Mar 2025 - Feb 2026
  What will be measured:
  The output is a single figure. We aim to depict a visual representation of the resources, key activities, outputs, outcomes, and plausible causal pathways connecting them.
Written programme description | Mar 2025 - Feb 2026
  What will be reported:
  The investigators will report the narrative detailed description of the programme.
  How will it be measured or reported: The frameworks used are TIDIER and AIMD.
Process indicators | Mar 2025 - Feb 2026
  What will be measured:
  Number of older adults with Clinical frailty scale (CFS) score 4-5, number of older adults who completed intrinsic capacity screening, number of older adults who actualised follow-up appointments.
  How will it be measured: Data collection will be from healthcare providers on the ground.
Fidelity of implementation strategy: Educational meetings, Part 1 | Mar 2025 - Feb 2026
  What will be measured:
  Actor: Who executed the educational meetings.
  How will it be measured: Data collection will be from healthcare providers on the ground.
Fidelity of implementation strategy: Educational meetings, Part 2 | Mar 2025 - Feb 2026
  What will be measured:
  Action target: Who attended the meetings
  How will it be measured: Data collection will be from healthcare providers on the ground.
Fidelity of implementation strategy: Educational meetings, Part 3 | Mar 2025 - Feb 2026
  What will be measured:
  Temporality: Frequency of meetings
  How will it be measured: Data collection will be from healthcare providers on the ground.
Fidelity of implementation strategy: Educational meetings, Part 4 | Mar 2025 - Feb 2026
  What will be measured:
  Dose: Number of meetings that each healthcare provider attended.
  How will it be measured: Data collection will be from healthcare providers on the ground.
Fidelity of implementation strategy: Educational meetings, Part 5 | Mar 2025 - Feb 2026
  What will be measured:
  Action: Content (topics)/style (lecture, didactic) of educational meetings
  How will it be measured: Data collection will be from healthcare providers on the ground.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Sum, PhD, Principal Investigator — Geriatric Education and Research Institute

IPD SHARING:
Plan to Share IPD: No
The information will not be shared due to confidentiality.

REFERENCES:
- [Background] O'Donovan MR, Sezgin D, Liew A, O'Caoimh R. Burden of disease, disability-adjusted life years and frailty prevalence. QJM. 2019 Apr 1;112(4):261-267. doi: 10.1093/qjmed/hcy291. PMID 30541151
- [Background] Milat A, Lee K, Conte K, Grunseit A, Wolfenden L, van Nassau F, Orr N, Sreeram P, Bauman A. Intervention Scalability Assessment Tool: A decision support tool for health policy makers and implementers. Health Res Policy Syst. 2020 Jan 3;18(1):1. doi: 10.1186/s12961-019-0494-2. PMID 31900230
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Sutton E, Catling J, Segaert K, Veldhuijzen van Zanten J. Cognitive Health Worries, Reduced Physical Activity and Fewer Social Interactions Negatively Impact Psychological Wellbeing in Older Adults During the COVID-19 Pandemic. Front Psychol. 2022 Feb 17;13:823089. doi: 10.3389/fpsyg.2022.823089. eCollection 2022. PMID 35250763
- [Background] Lopez-Teros T, Gutierrez-Robledo LM, Perez-Zepeda MU. Gait Speed and Handgrip Strength as Predictors of Incident Disability in Mexican Older Adults. J Frailty Aging. 2014;3(2):109-12. doi: 10.14283/jfa.2014.10. PMID 27049903
- [Background] Tan WS, Nai ZL, Tan HTR, Nicholas S, Choo R, Ginting ML, Tan E, Teng PHJ, Lim WS, Wong CH, Ding YY; Geriatric Services Hub Programme Group. Protocol for a mixed-methods and multi-site assessment of the implementation process and outcomes of a new community-based frailty programme. BMC Geriatr. 2022 Jul 15;22(1):586. doi: 10.1186/s12877-022-03254-6. PMID 35840898
- [Background] Grigor'ev EG, Pankratova VA, Cherkashin AF. [Case of severe combined trauma]. Khirurgiia (Mosk). 1979 Oct;(10):109-10. No abstract available. Russian. PMID 522389
- [Background] Tulloch AJ, Moore V. A randomized controlled trial of geriatric screening and surveillance in general practice. J R Coll Gen Pract. 1979 Dec;29(209):733-40. PMID 536982
- [Background] Hyzy M, Bond R, Mulvenna M, Bai L, Dix A, Leigh S, Hunt S. System Usability Scale Benchmarking for Digital Health Apps: Meta-analysis. JMIR Mhealth Uhealth. 2022 Aug 18;10(8):e37290. doi: 10.2196/37290. PMID 35980732
- [Background] Kwan YH, Yoon S, Tan CS, Tai BC, Tan WB, Phang JK, Tan NC, Tan CYL, Quah YL, Koot D, Teo HH, Low LL. EMPOWERing Patients With Diabetes Using Profiling and Targeted Feedbacks Delivered Through Smartphone App and Wearable (EMPOWER): Protocol for a Randomized Controlled Trial on Effectiveness and Implementation. Front Public Health. 2022 Feb 25;10:805856. doi: 10.3389/fpubh.2022.805856. eCollection 2022. PMID 35284389
- [Background] Tay LB, Chua MP, Tay EL, Chan HN, Mah SM, Latib A, Wong CQ, Ng YS. Multidomain Geriatric Screen and Physical Fitness Assessment Identify Prefrailty/Frailty and Potentially Modifiable Risk Factors in Community-Dwelling Older Adults. Ann Acad Med Singap. 2019 Jun;48(6):171-180. PMID 31377761
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Smith JD, Li DH, Rafferty MR. The Implementation Research Logic Model: a method for planning, executing, reporting, and synthesizing implementation projects. Implement Sci. 2020 Sep 25;15(1):84. doi: 10.1186/s13012-020-01041-8. PMID 32988389
- [Background] Pua YH, Tay L, Clark RA, Thumboo J, Tay EL, Mah SM, Ng YS. Screening accuracy of percentage predicted gait speed for prefrailty/frailty in community-dwelling older adults. Geriatr Gerontol Int. 2022 Aug;22(8):575-580. doi: 10.1111/ggi.14418. Epub 2022 Jun 18. PMID 35716008
- [Background] Pua YH, Tay L, Clark RA, Thumboo J, Tay EL, Mah SM, Ng YS. Reference Ranges for Gait Speed and Sit-to-Stand Performance in a Cohort of Mobility-Intact Community-Dwelling Older Adults From Singapore. J Am Med Dir Assoc. 2022 Sep;23(9):1579-1584.e1. doi: 10.1016/j.jamda.2021.12.045. Epub 2022 Feb 10. PMID 35151629
- [Background] Clark RA, Pua YH, Bower KJ, Bechard L, Hough E, Charlton PC, Mentiplay B. Validity of a low-cost laser with freely available software for improving measurement of walking and running speed. J Sci Med Sport. 2019 Feb;22(2):212-216. doi: 10.1016/j.jsams.2018.07.005. Epub 2018 Jul 17. PMID 30029889
- [Background] Van Damme J, Neiterman E, Oremus M, Lemmon K, Stolee P. Perspectives of older adults, caregivers, and healthcare providers on frailty screening: a qualitative study. BMC Geriatr. 2020 Feb 17;20(1):65. doi: 10.1186/s12877-020-1459-6. PMID 32066393
- [Background] Preston L, Chambers D, Campbell F, Cantrell A, Turner J, Goyder E. What evidence is there for the identification and management of frail older people in the emergency department? A systematic mapping review. Southampton (UK): NIHR Journals Library; 2018 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK493681/ PMID 29697231
- [Background] Dent E, Martin FC, Bergman H, Woo J, Romero-Ortuno R, Walston JD. Management of frailty: opportunities, challenges, and future directions. Lancet. 2019 Oct 12;394(10206):1376-1386. doi: 10.1016/S0140-6736(19)31785-4. PMID 31609229
- [Background] Welstead M, Luciano M, Russ TC, Muniz-Terrera G. Heterogeneity of Frailty Trajectories and Associated Factors in the Lothian Birth Cohort 1936. Gerontology. 2022;68(8):861-868. doi: 10.1159/000519240. Epub 2021 Sep 29. PMID 34587617
- [Background] Tanaka T, Takahashi K, Hirano H, Kikutani T, Watanabe Y, Ohara Y, Furuya H, Tetsuo T, Akishita M, Iijima K. Oral Frailty as a Risk Factor for Physical Frailty and Mortality in Community-Dwelling Elderly. J Gerontol A Biol Sci Med Sci. 2018 Nov 10;73(12):1661-1667. doi: 10.1093/gerona/glx225. PMID 29161342
- [Background] Fourteau M, Virecoulon Giudici K, Rolland Y, Vellas B, de Souto Barreto P. Associations Between Multidomain Lifestyle Interventions and Intrinsic Capacity Domains During Aging: A Narrative Review. JAR Life. 2020 Sep 3;9:16-25. doi: 10.14283/jarlife.2020.6. eCollection 2020. PMID 36922921
- [Background] Bevilacqua R, Soraci L, Stara V, Riccardi GR, Corsonello A, Pelliccioni G, Lattanzio F, Casaccia S, Moller J, Wieching R, Ogawa T, Watanabe S, Kokobun K, Kondo I, Takano E, Maranesi E. A systematic review of multidomain and lifestyle interventions to support the intrinsic capacity of the older population. Front Med (Lausanne). 2022 Jul 15;9:929261. doi: 10.3389/fmed.2022.929261. eCollection 2022. PMID 35911409
- [Background] Cameron ID, Fairhall N, Langron C, Lockwood K, Monaghan N, Aggar C, Sherrington C, Lord SR, Kurrle SE. A multifactorial interdisciplinary intervention reduces frailty in older people: randomized trial. BMC Med. 2013 Mar 11;11:65. doi: 10.1186/1741-7015-11-65. PMID 23497404
- [Background] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Background] Chew J, Lim JP, Yew S, Yeo A, Ismail NH, Ding YY, Lim WS. Disentangling the Relationship between Frailty and Intrinsic Capacity in Healthy Community-Dwelling Older Adults: A Cluster Analysis. J Nutr Health Aging. 2021;25(9):1112-1118. doi: 10.1007/s12603-021-1679-2. PMID 34725670
- [Background] Lim YJ, Ng YS, Sultana R, Tay EL, Mah SM, Chan CHN, Latib AB, Abu-Bakar HM, Ho JCY, Kwek THH, Tay L. Frailty Assessment in Community-Dwelling Older Adults: A Comparison of 3 Diagnostic Instruments. J Nutr Health Aging. 2020;24(6):582-590. doi: 10.1007/s12603-020-1396-2. PMID 32510110
- [Background] Yu R, Amuthavalli Thiyagarajan J, Leung J, Lu Z, Kwok T, Woo J. Validation of the Construct of Intrinsic Capacity in a Longitudinal Chinese Cohort. J Nutr Health Aging. 2021;25(6):808-815. doi: 10.1007/s12603-021-1637-z. PMID 34179938
- [Background] Zeng X, Shen S, Xu L, Wang Y, Yang Y, Chen L, Guan H, Zhang J, Chen X. The Impact of Intrinsic Capacity on Adverse Outcomes in Older Hospitalized Patients: A One-Year Follow-Up Study. Gerontology. 2021;67(3):267-275. doi: 10.1159/000512794. Epub 2021 Mar 18. PMID 33735899
- [Background] Belloni G, Cesari M. Frailty and Intrinsic Capacity: Two Distinct but Related Constructs. Front Med (Lausanne). 2019 Jun 18;6:133. doi: 10.3389/fmed.2019.00133. eCollection 2019. PMID 31275941
- [Background] Portegijs E, Rantakokko M, Viljanen A, Sipila S, Rantanen T. Identification of Older People at Risk of ADL Disability Using the Life-Space Assessment: A Longitudinal Cohort Study. J Am Med Dir Assoc. 2016 May 1;17(5):410-4. doi: 10.1016/j.jamda.2015.12.010. Epub 2016 Jan 21. PMID 26805752
- [Background] Portegijs E, Rantakokko M, Viljanen A, Sipila S, Rantanen T. Is frailty associated with life-space mobility and perceived autonomy in participation outdoors? A longitudinal study. Age Ageing. 2016 Jul;45(4):550-3. doi: 10.1093/ageing/afw072. Epub 2016 Apr 28. PMID 27126330
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Ma L, Chhetri JK, Zhang Y, Liu P, Chen Y, Li Y, Chan P. Integrated Care for Older People Screening Tool for Measuring Intrinsic Capacity: Preliminary Findings From ICOPE Pilot in China. Front Med (Lausanne). 2020 Nov 30;7:576079. doi: 10.3389/fmed.2020.576079. eCollection 2020. PMID 33330532
- [Background] Tavassoli N, de Souto Barreto P, Berbon C, Mathieu C, de Kerimel J, Lafont C, Takeda C, Carrie I, Piau A, Jouffrey T, Andrieu S, Nourhashemi F, Beard JR, Soto Martin ME, Vellas B. Implementation of the WHO integrated care for older people (ICOPE) programme in clinical practice: a prospective study. Lancet Healthy Longev. 2022 Jun;3(6):e394-e404. doi: 10.1016/S2666-7568(22)00097-6. Epub 2022 Jun 9. PMID 36098317
- [Background] Kojima G, Taniguchi Y, Iliffe S, Jivraj S, Walters K. Transitions between frailty states among community-dwelling older people: A systematic review and meta-analysis. Ageing Res Rev. 2019 Mar;50:81-88. doi: 10.1016/j.arr.2019.01.010. Epub 2019 Jan 16. PMID 30659942
- [Background] Liu S, Kang L, Liu X, Zhao S, Wang X, Li J, Jiang S. Trajectory and Correlation of Intrinsic Capacity and Frailty in a Beijing Elderly Community. Front Med (Lausanne). 2021 Dec 9;8:751586. doi: 10.3389/fmed.2021.751586. eCollection 2021. PMID 34957141
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Woodhouse L, Rodriguez-Manas L, Fried LP, Woo J, Aprahamian I, Sanford A, Lundy J, Landi F, Beilby J, Martin FC, Bauer JM, Ferrucci L, Merchant RA, Dong B, Arai H, Hoogendijk EO, Won CW, Abbatecola A, Cederholm T, Strandberg T, Gutierrez Robledo LM, Flicker L, Bhasin S, Aubertin-Leheudre M, Bischoff-Ferrari HA, Guralnik JM, Muscedere J, Pahor M, Ruiz J, Negm AM, Reginster JY, Waters DL, Vellas B. Physical Frailty: ICFSR International Clinical Practice Guidelines for Identification and Management. J Nutr Health Aging. 2019;23(9):771-787. doi: 10.1007/s12603-019-1273-z. PMID 31641726
- [Background] Gutierrez-Robledo LM, Garcia-Chanes RE, Gonzalez-Bautista E, Rosas-Carrasco O. Validation of Two Intrinsic Capacity Scales and Its Relationship with Frailty and Other Outcomes in Mexican Community-Dwelling Older Adults. J Nutr Health Aging. 2021;25(1):33-40. doi: 10.1007/s12603-020-1555-5. PMID 33367460
- [Background] Lee JQ, Ding YY, Latib A, et alINtrinsic Capacity and its RElAtionship With Life-SpacE Mobility (INCREASE): a cross-sectional study of community-dwelling older adults in SingaporeBMJ Open 2021;11:e054705. doi: 10.1136/bmjopen-2021-054705
- [Background] World Health Organization. The International Classification of functioning, disability and health. 1149. The International Classification of Functioning, Disability and Health 2002: 1-22
- [Background] Woo, J. Frailty, Successful Aging, Resilience, and Intrinsic Capacity: a Cross-disciplinary Discourse of the Aging Process. Curr Geri Rep 8, 67-71 (2019). https://doi.org/10.1007/s13670-019-0276-2
- [Background] Vermeiren S, Vella-Azzopardi R, Beckwee D, Habbig AK, Scafoglieri A, Jansen B, Bautmans I; Gerontopole Brussels Study group. Frailty and the Prediction of Negative Health Outcomes: A Meta-Analysis. J Am Med Dir Assoc. 2016 Dec 1;17(12):1163.e1-1163.e17. doi: 10.1016/j.jamda.2016.09.010. PMID 27886869
- [Background] Beard JR, Si Y, Liu Z, Chenoweth L, Hanewald K. Intrinsic Capacity: Validation of a New WHO Concept for Healthy Aging in a Longitudinal Chinese Study. J Gerontol A Biol Sci Med Sci. 2022 Jan 7;77(1):94-100. doi: 10.1093/gerona/glab226. PMID 34343305
- [Background] Tay L, Tay EL, Mah SM, Latib A, Koh C, Ng YS. Association of Intrinsic Capacity with Frailty, Physical Fitness and Adverse Health Outcomes in Community-Dwelling Older Adults. J Frailty Aging. 2023;12(1):7-15. doi: 10.14283/jfa.2022.28. PMID 36629078
- [Background] Liu S, Yu X, Wang X, Li J, Jiang S, Kang L, Liu X. Intrinsic Capacity predicts adverse outcomes using Integrated Care for Older People screening tool in a senior community in Beijing. Arch Gerontol Geriatr. 2021 May-Jun;94:104358. doi: 10.1016/j.archger.2021.104358. Epub 2021 Jan 28. No abstract available. PMID 33548677
- [Background] Beard JR, Jotheeswaran AT, Cesari M, Araujo de Carvalho I. The structure and predictive value of intrinsic capacity in a longitudinal study of ageing. BMJ Open. 2019 Nov 2;9(11):e026119. doi: 10.1136/bmjopen-2018-026119. PMID 31678933
- [Background] Cesari M, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Cooper C, Martin FC, Reginster JY, Vellas B, Beard JR. Evidence for the Domains Supporting the Construct of Intrinsic Capacity. J Gerontol A Biol Sci Med Sci. 2018 Nov 10;73(12):1653-1660. doi: 10.1093/gerona/gly011. PMID 29408961
- [Background] Beard JR, Officer AM, Cassels AK. The World Report on Ageing and Health. Gerontologist. 2016 Apr;56 Suppl 2:S163-6. doi: 10.1093/geront/gnw037. No abstract available. PMID 26994257
- [Background] Chen C, Lim JT, Chia NC, Wang L, Tysinger B, Zissimopolous J, Chong MZ, Wang Z, Koh GC, Yuan JM, Tan KB, Chia KS, Cook AR, Malhotra R, Chan A, Ma S, Ng TP, Koh WP, Goldman DP, Yoong J. The Long-Term Impact of Functional Disability on Hospitalization Spending in Singapore. J Econ Ageing. 2019;14:100193. doi: 10.1016/j.jeoa.2019.02.002. Epub 2019 Feb 27. PMID 31857943
- [Derived] Wang Q, Ginting ML, Ho E, Goh SF, Gao J, Tan WS, Ding YY, Ng WLD, Ng JCA, Kwek SC, Hui RJY, Wang ZS, Ng CJ, Sum G; IMPACTFrail Group. Development and Feasibility Assessment of an Intrinsic Capacity Program in Primary Care: Protocol for an Implementation Science Approach. JMIR Res Protoc. 2026 Feb 2;15:e84257. doi: 10.2196/84257. PMID 41628431
- See also: 1. Life expectancy at birth. Data based on the latest United Nations Population Division estimates. — https://www.worldometers.info/demographics/life-expectancy/
- See also: Brooke J. SUS: a quick and dirty usability scale. ResearchGate. 1995 — https://www.researchgate.net/publication/228593520_SUS_A_quick_and_dirty_usability_scale
- See also: WHO. Adherence to long term therapies: evidence for action. 2003. — https://apps.who.int/iris/handle/10665/42682
- See also: 59. Infocomm Media Development Authority. Annual survey on infocomm usagein households and by individuals for 2017. Singapore: Infocomm Media Development Authority 2018. — https://www.imda.gov.sg/-/media/Imda/Files/
- See also: Singapore survey finds elderly unreceptive to digital health services. Health IT News. July 2021 — https://www.healthcareitnews.com/news/asia/singapore-survey-finds-elderly-unreceptive-digital-health-services
- See also: Integrated care for older people. Implementation framework. Guidance for systems and services. World Health Organization — https://www.who.int/publications/i/item/9789241515993
- See also: Guidance on person-centred assessment and pathways in primary care. Handbook. World Health Organization — https://www.afro.who.int/publications/handbook-guidance-person-centred-assessment-and-pathways-primary-care
- See also: World Report on Ageing and Health. World Health Organization; 2015 — https://www.who.int/publications/i/item/9789241565042
- See also: WHO. Integrated care for older people (ICOPE) implementation programme: findings from the "ready" phase. — https://www.who.int/publications/i/item/9789240048355
- See also: WHO . Integrated care for older people: guidelines on community-level interventions to manage declines in intrinsic capacity. Geneva: World Health Organization 2017 — https://www.who.int/publications/i/item/9789241550109
- See also: WHO Clinical Consortium on Healthy Ageing. Report of consortium meeting 1-2 December 2016 in Geneva, Switzerland. Geneva: World Health Organization 2017 — https://www.who.int/publications/i/item/WHO-FWC-ALC-17.2